CLINICAL TRIAL: NCT02916914
Title: Impact of Feeding Interval of Preterms on the Time of Transition From Tube Feeding to Oral Feeding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Etlik Zubeyde Hanim Womens' Health and Teaching Hospital (Unknown)
Responsible Party: Principal Investigator, Sezin Unal, MD, Etlik Zubeyde Hanim Womens' Health and Teaching Hospital
Organization: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EZH/2015/4
Record Dates: First submitted 2016-09-08; First posted 2016-09-28 (Estimated); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Bottlefeeding; Infant, Premature, Diseases
Keywords: preterm; feeding; oral transition
MeSH Terms: conditions — Bottle Feeding; Infant, Premature, Diseases; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Q2 feeding (Other): feeding intervals: 2 hours
  Interventions: Other: Q2 feeding
- Q3feeding (No Intervention): feeding intervals: 3 hours

INTERVENTIONS:
Other: Q2 feeding — Infants are going to be fed every 2 hours
  Arms: Q2 feeding

SUMMARY:
Preterms are usually fed with intervals of either two or three hours during their stay in neonatal intensive care unit. Recommendations of World Health Organization about feeding regimens, 3-hourly for infants 1500 - 2000 gr, and 2-hourly for infants 1000 - 1500 gr, are not proposed with regards to results of randomized controlled trials. Investigators aimed to investigate the impact of 2-hourly feeding on time of transition from orogastric to oral feeding.

DETAILED DESCRIPTION:
Preterms are usually fed with intervals of either two or three hours during their stay in neonatal intensive care unit. Recommendations of World Health Organization about feeding regimens, 3-hourly for infants 1500 - 2000 gr, and 2-hourly for infants 1000 - 1500 gr, are not proposed with regards to results of randomized controlled trials.

Stomach volume of preterms varies a wide range of upto 20 ml. This should be taken into consideration during the process of feeding of preterms in neonatal intensive care unit. Trials were focused on early neonatal outcomes and it was found that duration of phototherapy and nasal noninvasive ventilation, and time to achieve full enteral feeds were shorter during 2-hourly feeding when compared to 3-hourly feeding, on the other hand 3-hourly feeding was shown to accelerate the stomach emptying. Besides, duration of catheterization, and ratio of feeding intolerance, apnea, and hypoglycemia were found to be similar infants who fed either 2 or 3-hourly.

Investigators aimed to investigate the impact of two feeding regimens, 2-hourly or 3-hourly, on time of transition from orogastric to oral feeding in preterms.

Patients and Methods: Preterms of birth weight less that 1500 gr and gestational age smaller than 32 weeks are going to be eligible for study if no congenital anomalies exist. Regarding current clinical protocol infants are fed every 2 hours until they weigh 1500 gr, and every 3 hours afterwards. At the day that the infants reach 1500 gr of body weight, a randomization will be performed in to two groups, Intervention group: Q2 interval (2-hourly feeding) or Control group: Q3 interval (3-hourly feeding), due to study protocol. Infants with inherited metabolic disorders, congenital anomalies, neonatal sepsis, and surgical diseases and the ones who fed with exclusively formula will be excluded.

After randomization infants will be followed until discharge. The type of feeding, volume of each feed, weight gain per week, feeding intolerance (abdominal distention, vomiting, apnea, newly onset or increase of oxygen treatment demand), day of first oral feeding, time of transition from orogastric tube to oral feeding, duration of hospitalization will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. birth weight <= 1500 gr gr
2. gestational age <= 32 weeks
3. postnatal age at randomization: between 7 - 90 days

Exclusion Criteria:

* congenital anomaly
* multi organ failure
* sepsis
* surgical pathology
* inherited metabolic diseases
* exclusively formula feeding

Ages: 7 Days to 90 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-09-30 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
time of transition from orogastric to oral feeding | From date of birth to date of transition from orogastric to oral feeding or date of death, which ever came first, will be assessed up to 44th post menstrual age (days of life)

SECONDARY OUTCOMES:
feeding intolerance after randomization; intolerance events per week until discharge | From date of randomization to date of discharge or date of death, which ever came first, will be assessed up to 44th post menstrual age
duration of hospitalization | From date of birth to date of discharge or date of death, which ever came first, will be assessed up to 44th post menstrual age, (days of life)
weight gain per week until discharge | From date of randomization to date of discharge or date of death, which ever came first, will be assessed up to 44th post menstrual age, (grams/kg/week)

CONTACTS AND LOCATIONS:
Overall Officials: Sezin Unal, MD, Principal Investigator — Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Locations (1):
- EtlikWHTH, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergman NJ. Neonatal stomach volume and physiology suggest feeding at 1-h intervals. Acta Paediatr. 2013 Aug;102(8):773-7. doi: 10.1111/apa.12291. Epub 2013 Jun 3. PMID 23662739
- [Background] Dhingra A, Agrawal SK, Kumar P, Narang A. A randomised controlled trial of two feeding schedules in neonates weighing <or=1750 g. J Matern Fetal Neonatal Med. 2009 Mar;22(3):198-203. doi: 10.1080/14767050802385749. PMID 19330703
- [Background] Rudiger M, Herrmann S, Schmalisch G, Wauer RR, Hammer H, Tschirch E. Comparison of 2-h versus 3-h enteral feeding in extremely low birth weight infants, commencing after birth. Acta Paediatr. 2008 Jun;97(6):764-9. doi: 10.1111/j.1651-2227.2008.00774.x. Epub 2008 Apr 16. PMID 18422805
- [Background] DeMauro SB, Abbasi S, Lorch S. The impact of feeding interval on feeding outcomes in very low birth-weight infants. J Perinatol. 2011 Jul;31(7):481-6. doi: 10.1038/jp.2010.153. Epub 2011 Jan 20. PMID 21252961